CLINICAL TRIAL: NCT02516826
Title: The Effect of Rosuvastatin and Olmesartan on the Progression of Coronary Atherosclerotic Disease by Smart Angioplasty Research Team: SMART-ROAD Trial
Brief Title: The Effect of Rosuvastatin and Olmesartan on the Progression of Coronary Atherosclerotic Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-01-055
Record Dates: First submitted 2015-08-04; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable | interventions — Rosuvastatin Calcium; olmesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rosuvastatin Arm (Experimental): Rosuvastatin 10mg in combination with placebo of Olmesartan 20mg plus placebo of Olmesartan/Rosuvastatin(Combination) 20/10mg orally once daily
  Interventions: Drug: Rosuvastatin; Drug: Placebo of Olmesartan; Drug: Placebo of Rosuvastatin/Olmesartan(Combination)
- Olmesartan Arm (Experimental): Olmesartan 20mg in combination with placebo of Rosuvastatin 10mg plus placebo of Olmesartan/Rosuvastatin(Combination) 20/10mg orally once daily
  Interventions: Drug: Olmesartan; Drug: Placebo of Rosuvastatin; Drug: Placebo of Rosuvastatin/Olmesartan(Combination)
- Combination Arm (Experimental): Olmesartan/Rosuvastatin(Combination) 20/10mg in combination with placebo of Rosuvastatin 10mg plus placebo of Olmesartan 20mg
  Interventions: Drug: Combination; Drug: Placebo of Rosuvastatin; Drug: Placebo of Olmesartan

INTERVENTIONS:
Drug: Rosuvastatin
  Arms: Rosuvastatin Arm
Drug: Olmesartan
  Arms: Olmesartan Arm
Drug: Combination — Rosuvastatin/Olmesartan(Combination)
  Arms: Combination Arm
Drug: Placebo of Rosuvastatin
  Arms: Combination Arm; Olmesartan Arm
Drug: Placebo of Olmesartan
  Arms: Combination Arm; Rosuvastatin Arm
Drug: Placebo of Rosuvastatin/Olmesartan(Combination)
  Arms: Olmesartan Arm; Rosuvastatin Arm

SUMMARY:
1. Stains have demonstrated consistent benefits to reduce cardiovascular events in several primary and secondary prevention trials. The suppression of plaque progression or regression may be a part of mechanism of clinical benefit. The intravascular ultrasound studies demonstrated that intensive statin therapy can regress or inhibit the progression of coronary atherosclerosis.
2. Unregulated renin-angiotensin system is important in the pathogenesis of cardiovascular disease. Angiotensin receptor antagonists (ARB) have been reported to improve clinical outcomes in patients with heart failure, left ventricular dysfunction, myocardial infarction, and high-risk patients. Several small studies showed that ARBs were effective to inhibit the progression of coronary atherosclerosis by intravascular ultrasound examination.
3. The combined therapy with statins and ARBs may be additive or synergistic effects on the atherosclerosis regression as well as to improve endothelial dysfunction and insulin resistance in addition to lowering cholesterol levels and blood pressure when compared with either monotherapy in patients.
4. Serial computed tomography angiography (CTA) can be utilized to assess the effect of treatment on coronary plaque morphology. In addition to the assessment of luminal stenosis, CTA also allows characterization of plaque morphology.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at 19 years~70 years of age
2. Patients undergoing coronary CTA with coronary artery stenosis 30~70%
3. Informed consent
4. Appropriate CT resolution enough to measure of plaque volume
5. Patients who are stain and renin-angiotensin system blocker naïve at least for 1 year

Exclusion Criteria:

1. Patients with>=70% luminal stenosis or requiring percutaneous coronary intervention(PCI)
2. Severely calcifiedcoronary artery
3. Patients who have a history of previous PCI or coronary artery bypass grafting surgery.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
PAV(nominal change of percent atheroma volume) in the proximal to mid segments of major epicardial coronary arteries | Over the 48weeks
  Left main, LAD proximal to mid (from ostium to a large second diagonal branch), LCX proximal (from ostium to a large first obtuse marginal branch), RCA (from ostium to a distal bifurcation)

SECONDARY OUTCOMES:
TAV (nominal change of total atheroma volume) in the proximal to mid segments of major epicardial coronary arteries | Over the 48weeks
  Left main, LAD proximal to mid (from ostium to a large second diagonal branch), LCX proximal (from ostium to a large first obtuse marginal branch), RCA (from ostium to a distal bifurcation)
LAPV (nominal change of percent low attenuation plaque volume) | Over the 48weeks
Nominal change of atheroma volume in 10 mm subsegment with greatest disease severity | Over the 48weeks
Change in insulin resistance | Over the 48weeks
Major adverse cardiac events | Over the 48weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, PhD, Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Cardiac and Vascular Center; Samsung Medical Center, Seoul, South Korea